CLINICAL TRIAL: NCT04847492
Title: Evaluation of Maxillary En-masse Retraction Rate Supported by Mini-screws and Assisted by Traditional or Flapless Corticotomy Techniques: A Randomized Controlled Trial
Brief Title: Evaluation of Upper Anterior Teeth Retraction Rate Assisted by Two Corticotomy Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-03-2021
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Class II Division 1 Malocclusion
Keywords: En-masse; retraction; corticotomy; flapless; miniscrew; upper anterior teeth
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional corticotomy (Active Comparator): Adult patients will be treated by en-masse retraction associated with traditional corticotomy.
  Interventions: Procedure: Traditional corticotomy
- Flapless corticotomy (Experimental): Adult patients will be treated by en-masse retraction associated with flapless corticotomy.
  Interventions: Procedure: Flapless corticotomy

INTERVENTIONS:
Procedure: Traditional corticotomy — A full-thickness mucoperiosteal flap will be elevated including the interdental papilla, and extended from the distal side of the second premolar on the right side to the same position on the left side without performing any vertical releasing incisions. Then, one vertical incision between the roots of upper anterior teeth and two vertical incisions in the site of first premolar extraction will be made by the piezosurgery knife.
  Arms: Traditional corticotomy
Procedure: Flapless corticotomy — Vertical soft-tissue incisions will be made on the buccal and palatal gingiva by using a blade N.15. One incision will be made between the roots of the six upper anterior teeth, and two incisions will be made between the upper canines and the second premolars.
  Arms: Flapless corticotomy

SUMMARY:
This study aims to assess the dental changes, periodontal health and the pulp vitality in mini-screw supported en-masse retraction associated with traditional or flapless corticotomy techniques.

40 adult patients exhibiting class II division 1 malocclusion requiring upper first premolar extractions followed by en-masse retraction will participate in the study. They will be randomly and equally distributed into two groups: traditional corticotomy (20 patients) versus flapless corticotomy (20 patients). The corticotomy procedure will be performed pre-retraction. The dental changes will be assessed using dental casts. The impressions will be taken after finishing the leveling and alignment phase and before starting the en-masse retraction (T0), 1 month (T1), 2 months (T2), 3 months (T3), 4 months (T4), and 5 months (T5) following the onset of en-masse retraction. The final impression will be considered at the end of the en-masse retraction (when the canines reach Class Ι relationship).

DETAILED DESCRIPTION:
One of the most important challenges in daily practice is prolonged orthodontic treatment duration. For that lots of therapeutic procedures have been introduced to minimize orthodontic treatment time such as surgical interventions. Even though the traditional corticotomy with flap elevation proved to be effective in accelerating different types of tooth movement, it has been deemed aggressive. Therefore, minimally invasive surgical techniques have been proposed and labeled 'flapless corticotomies'.

In flapless corticotomy group, vertical soft-tissue incisions will be made on the buccal and palatal gingiva by using a blade N.15. One incision will be made between the roots of the six upper anterior teeth, and two incisions will be made between the upper canines and second premolars. The incisions will be 5 mm long and started 4 mm apical to the interdental papilla. Then a piezosurgery knife will be inserted to perform the cortical alveolar incisions with 3-mm in-depth and 8-mm in length. No suturing will be needed.

In traditional corticotomy group, a full-thickness mucoperiosteal flap will be elevated including the interdental papilla, and extended from the distal side of the second premolar on the right side to the same position on the left side without performing any vertical releasing incisions. The full-thickness flap will be extended 3 mm above the root apices, from the buccal and palatal sides, knowing that the incision in the incisal papilla region will be done around it with a (V) or (U) shape. Then, one vertical incision between the roots of upper anterior teeth and two vertical incisions in the site of first premolar extraction will be made by the piezosurgery knife. The vertical incisions will be connected by a horizontal incision using the piezosurgery knives. The vertical incisions will be 3 mm in depth, starting 2-3 mm apical to the alveolar crest, and extending 3 mm beyond the root apices. The interrupted technique of suturing will be done using a non-absorbent 3-0 black silk.

The en-masse retraction will be begun 4 days after carrying out the corticotomy procedure using 0.019×0.025-inch SS archwires with 8-10-mm long soldered hooks located distal to the lateral incisors. NiTi closed coil springs with 9-mm long will be extended from the mini-screws to the soldered hooks and applied 250-g of force per side. The patients' follow-up appointments will be every 2 weeks. The force will be measured on every appointment and adjusted if needed. The endpoint of the monitoring period will be the session when canines reached a class Ι relationship.

ELIGIBILITY:
Inclusion Criteria:

1. Age range between 18 and 30 years.
2. Class II division 1 malocclusion requiring extraction of upper first premolars.
3. Mild to moderate skeletal class II malocclusion.
4. Normal or excessive anterior facial height.
5. No or mild crowding (tooth-size arch-length discrepancy ≤3 mm).
6. Overjet >5 mm and <10 mm.
7. Completion permanent dentition (regardless of third molars).
8. No previous orthodontic treatment.
9. No drug use or systematic disease that would affect the bone and tooth movement rate.
10. Healthy periodontium and good oral hygiene.

Exclusion Criteria:

1. Patients with previous orthodontic treatment.
2. Patients with severe skeletal dysplasia in all three dimensions.
3. Patients suffer from systemic diseases or syndromes
4. Patients on medication for systemic disorders, pregnancy or steroid therapy.
5. Patients showing any signs of active periodontal disease
6. Patients with severe crowding (≥ 3.5 mm) in maxillary arch
7. Patients with missing or extracted teeth in maxillary arch except third molar.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
The rate of en-masse retraction of upper anterior teeth. | The calculation of the rate of retraction will be done once the retraction procedures finish. It is expected to happen within 5 months
  The rate of en-masse retraction of upper anterior teeth (mm/month) in each group will be calculated.
  This outcome will be measured by the following steps:
  Drawing a projection from the upper canine apex to the middle palatal bone line.
  Drawing a projection from the upper central incisor edge to the middle palatal bone line.
  Drawing a projection from the mesial ending of the third palatal rugae to the middle palatal bone line.
  Measuring the distance (mm) between the canine apex and third palatal rugae projections.
  Measuring the distance (mm) between the central incisor edge and third palatal rugae projections.
  The rate of en-masse retraction will be measured by dividing the distance between the canine apex/central incisor edge projections and the third palatal rugae projection by the time elapsed between assessment times.
Change in the anteroposterior movement of the molar at 5 months | T0:1 day before the beginning of the retraction phase. T1: after 1 month of the beginning of retraction phase . T2: after 2 months. T3: after 3 months. T4: after 4 months. T5: immediately after the end of retraction phase (expected to be after 5 months)
  The anteroposterior movement of the molar (mm/month) in each group will be calculated.
  This outcome will be measured on the dental casts by drawing two projections from the central groove of the first maxillary molar and the mesial ending of the third palatal rugae to the middle palatal bone line. The anteroposterior movement of the first maxillary molar (mm) will be measured by dividing the distance between the two projections by the time elapsed between assessment times.
Change in the inter-canine width at 5 months | T0:1 day before the beginning of the retraction phase. T1: after 1 month of the beginning of retraction phase . T2: after 2 months. T3: after 3 months. T4: after 4 months. T5: immediately after the end of retraction phase (expected to be after 5 months)
  The change in the inter-canine width (mm/month) in each group will be calculated.
  Assessment will be performed by measuring the distance between the cusp tips of the two upper canines. This variable will be measured on dental casts.
Change in the inter-molar width at 5 months | T0:1 day before the beginning of the retraction phase. T1: after 1 month of the beginning of retraction phase . T2: after 2 months. T3: after 3 months. T4: after 4 months. T5: immediately after the end of retraction phase (expected to be after 5 months)
  The change in the inter-molar width (mm/month) in each group will be calculated.
  Assessment will be performed by measuring the distance between the the central groove of the two first maxillary molars. This variable will be measured on dental casts.

SECONDARY OUTCOMES:
The change in dental plaque index according to Silness and Loe | T0: immediately before the start of treatment; T1: one day before the commencement of the retraction phase; T2: immediately after the end of retraction phase (expected to be after 5 months)
  Assessment will be performed using a gingival probe. (0) = No plaque.
  1. = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  2. = Moderate accumulation of soft deposits within the gingival pocket, or on the tooth and gingival margin which can be seen with the naked eye.
  3. = Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
The change in gingival index according to Silness and Loe | T0: immediately before the start of treatment; T1: one day before the commencement of the retraction phase; T2: immediately after the end of retraction phase (expected to be after 5 months)
  Assessment will be performed using a gingival probe. (0) = Normal gingiva.
  1. = Mild inflammation: slight change in color, slight oedema. No bleeding on probing.
  2. = Moderate inflammation: redness, oedema and glazing. Bleeding on probing.
  3. = Sever inflammation: marked redness and oedema, ulceration, and tendency to spontaneous bleeding
The change in papillary bleeding index according to Muhlemann | T0: immediately before the start of treatment; T1: one day before the commencement of the retraction phase; T2: immediately after the end of retraction phase (expected to be after 5 months)
  Assessment will be performed using a gingival probe. (0) = No bleeding.
  1. = A single discreet bleeding point appears.
  2. = Several isolated bleeding points or a single fine line of blood appears.
  3. = The interdental triangle fills with blood shortly after probing.
  4. = Profuse bleeding occurs after probing; blood flows immediately into the marginal sulcus.
The change in gingival recession index according to Miller | T0: immediately before the start of treatment; T1: one day before the commencement of the retraction phase; T2: immediately after the end of retraction phase (expected to be after 5 months)
  The presence of gingival recession on the studied teeth was determined by using a gingival probe and naked eye view, with direct clinical measurement from the cemento-enamel junction to the edge of the free gingiva in the event of the recession.
Tooth vitality | T0: immediately before the start of treatment; T1: one day before the commencement of the retraction phase; T2: immediately after the end of retraction phase (expected to be after 5 months)
  Assessment will be performed from the maxillary right first molar to the maxillary left first molar by using Ethyl chloride spray (endo ice) at a temperature -50°.
  Each tooth will be subjected to this ice and the resultant outcome is dichotomous (the tooth is vital, the tooth is not vital).

CONTACTS AND LOCATIONS:
Overall Officials: Hanin Nizar Khlef, DDS,MSc, Principal Investigator — Specialist and Clinical Lecturer, Department of Orthodontics, University of Damascus; Mohammad Y Hajeer, DDS,MSc,PhD, Study Chair — Associate Professor of Orthodontics, University of Damascus Dental School, Damascus, Syria; Omar Heshmeh, DDS,MSc,PhD, Study Director — Professor of Oral and Maxillofacial Surgery, University of Damascus Dental School, Damascus, Syria
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Sibaie S, Hajeer MY. Assessment of changes following en-masse retraction with mini-implants anchorage compared to two-step retraction with conventional anchorage in patients with class II division 1 malocclusion: a randomized controlled trial. Eur J Orthod. 2014 Jun;36(3):275-83. doi: 10.1093/ejo/cjt046. Epub 2013 Jun 20. PMID 23787192
- [Background] Khlef HN, Hajeer MY, Ajaj MA, Heshmeh O. En-masse Retraction of Upper Anterior Teeth in Adult Patients with Maxillary or Bimaxillary Dentoalveolar Protrusion: A Systematic Review and Meta-analysis. J Contemp Dent Pract. 2019 Jan 1;20(1):113-127. PMID 31058623
- [Background] Alfawal AM, Hajeer MY, Ajaj MA, Hamadah O, Brad B. Effectiveness of minimally invasive surgical procedures in the acceleration of tooth movement: a systematic review and meta-analysis. Prog Orthod. 2016 Dec;17(1):33. doi: 10.1186/s40510-016-0146-9. Epub 2016 Oct 24. PMID 27696311
- [Background] Alfawal AMH, Hajeer MY, Ajaj MA, Hamadah O, Brad B. Evaluation of piezocision and laser-assisted flapless corticotomy in the acceleration of canine retraction: a randomized controlled trial. Head Face Med. 2018 Feb 17;14(1):4. doi: 10.1186/s13005-018-0161-9. PMID 29454369
- [Background] Khlef HN, Hajeer MY, Ajaj MA, Heshmeh O, Youssef N, Mahaini L. The effectiveness of traditional corticotomy vs flapless corticotomy in miniscrew-supported en-masse retraction of maxillary anterior teeth in patients with Class II Division 1 malocclusion: A single-centered, randomized controlled clinical trial. Am J Orthod Dentofacial Orthop. 2020 Dec;158(6):e111-e120. doi: 10.1016/j.ajodo.2020.08.008. Epub 2020 Nov 4. PMID 33158633
- [Derived] Khlef HN, Hajeer MY. Is It Possible to Achieve Favorable Accelerated Dental Changes with No Periodontal Complications When Retracting Upper Anterior Teeth Assisted by Flapless Corticotomy Compared to Traditional Corticotomy? A Two-Arm Randomized Controlled Trial. ScientificWorldJournal. 2022 Mar 7;2022:4261248. doi: 10.1155/2022/4261248. eCollection 2022. PMID 35295761